CLINICAL TRIAL: NCT01883895
Title: Exercise-induced Hypoalgesia After Comparative Forms of Anaerobic Training in Healthy Adults
Brief Title: Exercise-induced Hypoalgesia After Comparative Forms of Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0805
Record Dates: First submitted 2013-06-12; First posted 2013-06-21 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: Pain; exercise-induced hypoalgesia
MeSH Terms: conditions — Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: three treatment design, all participants will perform two exercise sessions (isometric exercise, concentric exercise), as well as a control session in a randomized manner. (This is not a cross-over design as each participant will have their own randomized order of sessions of exercise & control sessions.)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise treatment (Other): Concentric exercise: subject will utilize a dumbbell with elbow flexion exercise.
  Isometric exercise: Subjects will perform 5 sets of sustained muscle contraction.
  Control: Subjects will undergo a control arm where they will rest for approximately 10 minutes.
  Pain testing conducted by Forgionei-Barber pressure pain-stimulator for both the control and exercise treatments.
  Interventions: Device: Forgionei-Barber pressure-pain stimulator; Other: Concentric Exercise; Other: isometric exercise

INTERVENTIONS:
Device: Forgionei-Barber pressure-pain stimulator — Pain testing will be conducted using a Forgioni-Barber pressure-pain stimulator to deliver 3000-gm force to the middle digit of the non-dominant middle finger for up to 120 seconds. During stimulation, subjects will press a button attached to a timer when the pressure stimulus first becomes painful (pain threshold) and will also rate their perceived pain intensity using a 0-100 numeric pain rating scale at 20 second intervals during the 2 minute exposure to the pressure stimulus. This validated protocol has been used in previous research by investigators in this study. This will be used for both exercise sessions and the control session. Forgionei-Barber pressure-pain stimulator will be used.
Other: Concentric Exercise — Concentric testing will utilize a dumbbell with elbow flexion exercise. Subjects will perform 5 sets of 20 reps at 30% MVC. Pain testing will be conducted using a Forgionei-Barber pressure-pain stimulator immediately before and after the exercise.
Other: isometric exercise — When undergoing isometric exercise, subjects will perform 5 sets of sustained muscle contraction for 65 seconds using a hand-grip dynamometer. Pain testing will be conducted using a Forgionei-Barber pressure-pain stimulator immediately before and after the exercise.

SUMMARY:
The study involves recording response to discomfort following different forms of exercise. We think that there will be a increased pain tolerance following exercise but are unsure if there will be a difference between exercises.

DETAILED DESCRIPTION:
Known changes of the hypothalamic-pituitary-adrenal (HPA) axis, as well as other neurotransmitter systems, lead to alteration of peripheral and central nociception during acute and chronic stress. Exercise is one example of such physiologic stress. Exercise, in various forms, has been shown to exert effects on pain attenuation. Several studies have demonstrated post-exercise reduction in pain ratings, increased pain threshold as well as attenuation of pain-related increases in motor evoked potentials. This phenomenon is referred to as exercise-induced analgesia (EIA) or, perhaps more accurately, exercise-induced hypoalgesia (EIH).

Exercise at higher intensities and longer durations have the most robust evidence supporting their role in EIH. This is true of both long-duration aerobic training as well as high-intensity anaerobic training. This type of activity, however, may not be the most practical type of activity prescribed in a clinical population, especially in people with painful conditions, due to decreased conditioning and tolerance. Beyond long-duration and/or high-intensity aerobic exercise, there is growing evidence supporting the use of other forms and intensities of exercise that may induce EIH. Alternative forms of exercise, such as isometric stabilization, have been shown to decrease pain in a population of patients with low back pain. Koltyn and Arbogast investigated acute effects of exercise on pain perception and found that a single bout of resistance exercise at 75% of maximum intensity produces significant increases in pain thresholds and reductions in pain ratings.11 EIH can also occur during and following short duration (e.g., 1.5-5 min) and lower intensity (e.g., 15-50% max) isometric exercise. Along with high-intensity training, long-duration/low-intensity isometric contractions also have been found to produce an analgesic response. Studies have suggested different post-exercise pain responses in chronic pain populations compared to healthy controls, however questions still remain over the influence of various exercise intensities, protocols or types of contractions. Slater, et al examined the effects of eccentric exercise versus combined concentric-eccentric exercise at an intensity of 30% of max voluntary contraction (MVC) showed a significant increase in pain thresholds for both exercise protocols. Their study highlighted the need for further research to examine if changes also occur in response to single exercise modes. To date, no studies have compared EIH produced by isometric and concentric exercises at similar intensities and duration. Furthermore, little research in EIH has compared various forms of exercise to non-exercising controls.

Similar to EIH induced by aerobic exercise, the relationship of anaerobic exercise with hypoalgesia indicates a common mechanism that may be related to the augmentation of the central and peripheral nervous system through modulation of descending inhibition as well as the release of pain-relieving substances. There is possibly an orchestra of overlying and inter-related physiologic, social and psychologic mechanisms that contribute to hypoalgesia response to exercise. Because of confounding effect of various processes of all of these possible processes, it is important to evaluate specific exercise regimens that may provide most pain relief within the context of clinical practice. Although there is good evidence that long-duration aerobic, and high-intensity exercises modulate pain, these strategies may be difficult to apply in a clinical setting due to the disabling nature of painful conditions. Patients with such conditions may be more apt to comply with shorter duration exercises at lesser intensity. No studies to date have specifically addressed differences in pain response when comparing the EIH following anaerobic exercises using concentric and isometric training bouts as well as to a non-exercising control condition. Investigation of EIH in this study will improve understanding of nociceptive changes following therapeutic exercises in a clinical setting.

Aim 1: To examine changes in pain following two different types of exercise (isometric versus concentric contractions).

Hypothesis 1a: Pain will be significantly lower following both types of exercise in comparison to the non-exercising control condition. Currently, it is unclear whether pain responses will differ between the two exercise conditions since no previous research has been conducted in this area.

Aim 2: To examine whether men and women differ in pain responses following each exercise type.

Hypothesis 2: There will be no sex differences in the EIH responses.

We propose testing for EIH in healthy subjects by measuring potential differences in pressure pain intensity ratings with isometric versus concentric contractions as well as a control condition. This study seeks to determine if each of the two exercises produce EIH to same extent or are there differences in hypoalgesic response.

Primary outcomes: Pain intensity ratings: Subjects will rate pain intensity using a 0 (no pain) to 100 (most intense pain imaginable) pain rating scale before and after application of a validated pressure stimulator immediately prior to, and after exercise.

Secondary outcomes: Pain thresholds: Subjects will press a button attached to a timer out of view of the subject when the pressure stimulus first becomes painful. This will utilize a protocol recognized as a validated measurement of pain threshold.

We aim to examine the effect of exercise-induced hypoalgesia in healthy subjects. We will utilize a three-treatment randomized design where all subjects will undergo two exercise protocols as well as a control protocol on different dates. In order to essentially eliminate carry-over effect, we have elected to use a washout period of >48h to ensure adequate time for relief of any muscle pain or fatigue.

Subjects will first be tested for their one repetition voluntary maximum contraction (MVC) for the type of exercise being tested that day. Subjects will then be allowed to rest for 10-15 minutes while we review with them the exercise protocol and have them fill out questionnaires including demographics, State-Trait Anxiety Inventory and Pain Catastrophizing Scale. Immediately prior to exercise testing, we will record baseline pulse rate and blood pressure readings. Pain ratings and thresholds for pressure stimuli, as described below, will then be measured.

Subjects will then begin the exercise trial. Testing will be randomized so that subjects will perform protocols of either; a non-exercising control, concentric exercise or isometric exercise testing using all possible treatment sequences. Stratification for random sampling will be done using a block randomization scheme. For concentric testing, subjects will perform 5 sets of 20 reps at 30% MVC. When undergoing isometric exercise, subjects will perform 5 sets of sustained muscle contraction using the same duration of time it took to complete one set of 20 reps (as determined in pilot studies prior to initiation of this study). There will be a one-minute rest period between sets. Concentric testing will utilize a dumbbell with elbow flexion exercise. Isometric testing will be performed using a hand-grip dynamometer. Each exercise will be performed with the dominant arm/hand. Following exercise, subjects will also rate their perceived exertion and perceived muscle pain using the Borg Scale and Cook Scale, respectively. These are widely accepted and validated measures of perceived exertion and muscle pain. The control condition will consist of quiet rest for the same duration as the exercise conditions. At the end of the session, subjects will fill out two questionnaires: the State-Trait Anxiety Inventory and Situational Catastrophizing Scale. The validated questionnaires chosen to be completed at intake and post-testing will help to identify any confounding emotional or behavioral traits that may influence pain threshold and ratings.

Pain testing will be conducted using a Forgioni-Barber pressure-pain stimulator to deliver 3000-gm force to the middle digit of the non-dominant middle finger for up to 120 seconds. During stimulation, subjects will press a button attached to a timer when the pressure stimulus first becomes painful (pain threshold) and will also rate their perceived pain intensity using a 0-100 numeric pain rating scale at 20 second intervals during the 2 minute exposure to the pressure stimulus. This validated protocol has been used in previous research by investigators in this study.

Risks:

Subjects will insert the middle forefinger into the chute of the Forgioni-Barber pain stimulator where a non-fixed Lucite edge will contact the finger with a constant application of pressure from a 3 kg weight. This device creates a stimulus that is easy to apply and produces a distinct pain sensation with rapid onset and offset. It produces no tissue damage or psychological or physical health risk, and the subject is able to stop the stimulus at any time. The pain intensity is repeatable and readily discriminable throughout the stimulus application. Previous research has demonstrated that the Forgioni-Barber pressure-pain stimulator device, using the described procedure, is a safe device that produces a painful stimulus but does not cause tissue damage or injury. No significant adverse or side effects have been experienced or are expected from the exercise or pain stimulus. Temporary discomfort is expected during application of the pain stimulus, however this should resolve upon removal of the stimulus. There are no permanent consequences expected of this testing procedure. If the subject experiences excessive discomfort at any time during pain testing, we will immediately remove the stimulus. The subjects may withdraw from testing at any time during the research.

With exercise, there is a slight risk of muscle soreness or strain. We will mitigate risk of muscle strain by instructing the subjects to stop the exercise if they feel they are over-straining or begin to feel discomfort when performing the activity. The investigators will also be immediately available to assist, if needed, if the subject experiences discomfort during the exercise session. It is well known that repetitive contractions have a possibility of inducing delayed onset muscle soreness (DOMS). This is known to occur most often with eccentric exercises. Previous research has shown that there was no effect from DOMS using the intended protocol described and that a washout period of 24 hours was adequate with eccentric loading.

32 healthy normotensive males and females in the age range 18 to 40 years will be recruited from the community.

ELIGIBILITY:
Inclusion Criteria:

* normotensive
* age range 18 to 40 years

Exclusion Criteria:

* currently taking prescription medications
* current use of tobacco or recreational drugs including opiates and/or marijuana
* any chronic illness such as diabetes, cancer, fibromyalgia, or hypertension
* upper limb musculoskeletal pain, injury, or surgery that will limit ability to exercise

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nalini Sehgal, MD, Principal Investigator — University of Wisconsin Dept Ortho/Rehab; ben rawson, DO, Study Director — University of Wisconsin Dept Ortho/Rehab
Locations (1):
- University of Wisconsin Hospitals and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD with any other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Treatment: Concentric exercise will utilize a dumbbell with elbow flexion exercise. Isometric exercise will consist of submaximal exercise by squeezing the hand dynamometer with dominant hand at 30% of maximum for same duration as for concentric contractions,.
  Forgioni-Barber pressure-pain stimulator: Pain testing will be conducted using a Forgioni-Barber pressure-pain stimulator to deliver 3000-gm force to the middle digit of the non-dominant middle finger for up to 120 seconds. During stimulation, subjects will press a button attached to a timer when the pressure stimulus first becomes painful (pain threshold) and will also rate their perceived pain intensity using a 0-100 numeric pain rating scale at 20 second intervals during the 2 minute exposure to the pressure stimulus. This validated protocol has been used in previous research by investigators in this study.
  .
Period: Overall Study
Arm/Group | Exercise Treatment
Started | 34
Completed | 32
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 32 subjects completed study
  1 subject enrolled, but did not complete any treatments
  1 subject enrolled, but only completed the control session 33 baseline, and 1 drop-out = 34 total
Arm/Group | Exercise Treatment
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants] — Population: one subject did not complete and not included in analysis
  Participants
    number analyzed (Participants) | 32
    <=18 years | 0
    Between 18 and 65 years | 32
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: one subject did not complete and not included in analysis
  Participants
    number analyzed (Participants) | 32
    Female | 16
    Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: one subject did not complete and not included in analysis
  Participants
    number analyzed (Participants) | 32
    Hispanic or Latino | 1
    Not Hispanic or Latino | 31
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: one subject did not complete and not included in analysis
  Participants
    number analyzed (Participants) | 32
    American Indian or Alaska Native | 1
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 1
    White | 24
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity Ratings (0-100 Pain Scale)
Description: Subjects will rate pain intensity using a 0 (no pain) to 100 (most intense pain imaginable) pain rating scale before and after application of a validated pressure stimulator immediately prior to, and after exercise.
  Ratings will be recorded at 20 second intervals following each administration of the pressure stimulator for a total of 120 seconds. The ratings will then be averaged over all the time points.
Time Frame: Average pain rating over 120 seconds
Population: Participants completing both exercise sessions and control session
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Exercise Treatment: Concentric exercise: subject will utilize a dumbbell with elbow flexion exercise.
  Isometric exercise: Subjects will perform 5 sets of sustained muscle contraction.
  Control: Subjects will undergo a control arm where they will rest for approximately 10 minutes.
  Pain testing conducted Forgionei-Barber pressure pain stimulator
Arm/Group | Exercise Treatment
Number analyzed (Participants) | 32
scores on a scale
  control | 33.5 [22.7 to 44.5]
  concentric | 46.2 [31.3 to 61.1]
  isometric | 40.2 [31 to 60.9]

2. Secondary Outcome: Pain Threshold
Description: Subjects will press a button attached to a timer out of view of the subject when the pressure stimulus first becomes painful. This will utilize a protocol recognized as a validated measurement of pain threshold.
Time Frame: We will monitor the subject's reported pain thresholds during the two minute interval that the pressure stimulus is applied. Expected average is less than one minute.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise Treatment
Number analyzed (Participants) | 32
seconds
  control | 34.6 [16.4 to 52.7]
  concentric | 23.6 [-3.9 to 54.2]
  isometric | 24.5 [-4.5 to 53.5]

ADVERSE EVENTS:
Time Frame: All participants were tested over a 3 month period and adverse events were collected.
Arm/Group | Exercise Treatment
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes